CLINICAL TRIAL: NCT02081547
Title: IPC Status as a Surgical Quality Marker in Rectal Cancer Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: IPC
Record Dates: First submitted 2012-10-11; First posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Rectal Cancer
Keywords: rectal carcinoma; recurrence; pathology; cytology; free cancer cells; survival
MeSH Terms: conditions — Rectal Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 250 ml NaCl is poured in the abdominal cavity 3 times during the operation and is collected for accurence of cancer cells with Haemathoxylin&Eosin staining and immunohistochemistry. DNA sequencing is not performed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IPC status: presence of cancer cells.

SUMMARY:
Risk of local recurrence after rectal surgery is nationally 8% after curative surgery to 5%. Local recurrence rate after curative surgery varies between 3-7% in the variety of regions in the country. It is well known that the surgical technique total mesorectal excision (TME) has led to improved prognosis after rectal cancer surgery. TME surgery is difficult to perform and different factors affect the quality of TME preparations. Injuries in mesorectal fascia has been reported in up to 20% of patients who underwent TME surgery and most surgeons agree that this may be important for recurrences. However, it is unclear to what extent a damaged mesorectal fascia can be related to a worsening of prognosis in patients with rectal cancer.

Adjuvant oncological treatment in form of chemotherapy after surgery, is offers patients with unfavorable tumors based on the pathological examination. Patients with favorable tumors (less advanced) are not offered chemotherapy, even if the surgical technique was not optimal, ie. that there is damage in the mesorectal fascia, as evidence for this is lacking.

The presence of intraperitoneal cancer cells (IPC) is related to histopathological tumor stage of colorectal cancer. Incidence of IPC of intraperitoneal tumors (rectal cancer patients with tumors below the peritoneal reflection) is unclear.

Assessment of IPC status with cytology and immunohistochemistry is technically easy and could after TME surgery identify those patients who have an increased risk of tumor recurrence. In a positive IPC status, the patient would possibly benefit from either postoperative radiotherapy if the patient did not receive preoperative therapy, or postoperative oncological chemotherapy.

Tumour cells may be lysed in sterile water, and some surgeons rinse the abdominal cavity and the bowel distally to the tumour. Neither rinsing the abdomen or rectum in colorectal cancer is routinely occurring and the clinical benefit has not been established. The value of rinsing the abdomen after TME-surgery could also be studied by IPC status.

The study hypothesis is that the IPC status is dependent on the surgical quality of the specimen after TME-surgery in rectal cancer patients, and its presence leads to increased risk of local recurrence.

ELIGIBILITY:
Inclusion Criteria:

* rectal cancer patients that are going to be operated with bowel resection
* control patients (10 patients) - patients with different conditions that are going to be operated.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients with rectal cancer and 10 patients without rectal cancer that are operated.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-03 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
IPC status | One year
  Occurence of cancer cells per 100 mesothelial cell for the sample taken at the start of the surgery (sample 1). After completion of the TME-Surgery (sample 2) and after rinsing the abdomen (sample 3).
  The outcome will be assessed and presented when all patients are included (approximately dec 2013).

SECONDARY OUTCOMES:
TME quality | Day 1
  The surgeon grades the mesorectal completeness in a four grade scale.
local recurrence | 3-5 years after operation
  occurence of local recurrence.
Survival | after 3-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Maziar Hosseinali khani, MD PhD, Principal Investigator
Locations (2):
- Sweden (2):
  - Mälarsjukhuset Eskilstuna, Eskilstuna
  - Västmanlands sjukhus, Västerås

REFERENCES:
- [Result] Skipper D, Cooper AJ, Marston JE, Taylor I. Exfoliated cells and in vitro growth in colorectal cancer. Br J Surg. 1987 Nov;74(11):1049-52. doi: 10.1002/bjs.1800741130. PMID 3690235
- [Result] Kristensen AT, Wiig JN, Larsen SG, Giercksky KE, Ekstrom PO. Molecular detection (k-ras) of exfoliated tumour cells in the pelvis is a prognostic factor after resection of rectal cancer? BMC Cancer. 2008 Jul 27;8:213. doi: 10.1186/1471-2407-8-213. PMID 18655729
- [Result] Uras C, Altinkaya E, Yardimci H, Goksel S, Yavuz N, Kaptanoglu L, Akcal T. Peritoneal cytology in the determination of free tumour cells within the abdomen in colon cancer. Surg Oncol. 1996 Oct-Dec;5(5-6):259-63. doi: 10.1016/s0960-7404(96)80030-2. PMID 9129139
- [Result] Maeda K, Maruta M, Hanai T, Sato H, Horibe Y. Irrigation volume determines the efficacy of "rectal washout". Dis Colon Rectum. 2004 Oct;47(10):1706-10. doi: 10.1007/s10350-004-0659-z. PMID 15540303
- [Result] Noura S, Ohue M, Seki Y, Yano M, Ishikawa O, Kameyama M. Long-term prognostic value of conventional peritoneal lavage cytology in patients undergoing curative colorectal cancer resection. Dis Colon Rectum. 2009 Jul;52(7):1312-20. doi: 10.1007/DCR.0b013e3181a745a4. PMID 19571710